CLINICAL TRIAL: NCT02174887
Title: A Unicentric, Open Label, Mechanism of Action Trial, on the Biological Effect of Nab-paclitaxel Combined to Gemcitabine, in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Biological Effect of Nab-paclitaxel Combined to Gemcitabine in Metastatic Pancreatic Cancer
Acronym: MOAnab1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOAnab1-IPC 2012-010
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic adenocarcinoma; liver metastases
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-paclitaxel + Gemcitabine (Experimental): Gemcitabine 1 g/m² IV infusion over 30 minutes at D1-D8-D15 every 28 days in combination with Nab-paclitaxel 125 mg/m² IV infusion over 30 minutes at D1-D8-D15 every 28 days The patients will receive 2 cycles of treatment every 28 days
  Interventions: Drug: Nab-paclitaxel + Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel + Gemcitabine — Gemcitabine 1 g/m² IV infusion over 30 minutes at D1-D8-D15 every 28 days in combination with Nab-paclitaxel 125 mg/m² IV infusion over 30 minutes at D1-D8-D15 every 28 days
  The patients will receive 2 cycles of treatment every 28 days:

SUMMARY:
The prognostic of metastatic pancreatic adenocarcinoma is dismal and the treatment gold standard since the end of the 90s' is gemcitabine; unfortunately all trials testing combinations of gemcitabine with chemotherapeutic agents or targeted agents had failed to demonstrate any superiority over gemcitabine monotherapy.

In a recently published phase I/II study of combination of gemcitabine plus nab-paclitaxel in patients with metastatic pancreatic adenocarcinoma (PAC), the combination gave an impressive response rate of 48% (Gemcitabine 1g/m² and nab-paclitaxel 125 mg/m² once a week for 3 weeks, every 4 weeks). The safety profile was correct (fatigue, sensory neuropathy, nausea, haematological side effects). This efficacy can be related to an improvement of gemcitabine delivery to the tumor bed, as shown on preclinical studies: the response rate in xenografts was better with the combination; this improvement was associated with an increase of intratumoral gemcitabine concentration in mice receiving the combination when compared to mice receiving gemcitabine alone. This might be associated to modifications of peritumoral stroma with reduction of stromal content and increase in dilated vessels.

The aim of this study is to evaluate if the combination of nab-paclitaxel plus gemcitabine induces a modification in vascularization of pancreatic adenocarcinoma on the primary tumor and of liver metastases after 2 cycles of treatment by comparison to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Suspicion of pancreatic adenocarcinoma
3. With liver measurable metastases
4. Primary tumor non resected
5. First line systemic treatment
6. Correct haematological parameters
7. Adequate Blood chemistry levels
8. Life expectancy ≥ 2 months
9. PS: 0 - 2
10. Affiliation to French National social security or beneficiary
11. Signed informed consent.
12. Female patients must be surgically sterile, or be postmenopausal, or must commit to using reliable and appropriate methods of contraception during the study and during at least three months after the end of study treatment. All female patients with reproductive potential must have a negative pregnancy test (β HCG) within 72 hours prior to starting abraxane treatment. Breastfeeding is not allowed. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least six months after the end of the study treatment,

Exclusion Criteria:

1. Previous radiotherapy of the tumor
2. Patient has only locally advanced disease.
3. Previous treatment with gemcitabine
4. Active infection or severe concomitant disease
5. Serious Peripheral neuropathy
6. Known hypersensitivity or contraindication to any component of study drug formulation.
7. Pregnant or breastfeeding women
8. Other experimental treatment
9. History of malignancy in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
10. Known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
11. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity
12. Patient with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary, Hypersensitivity pneumonitis or multiple allergies
13. Patient uses Coumadin
14. Legal incapacity or limited legal capacity. Medical or psychological conditions not allowing the subject to complete the study or sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Vascularization parameters of pancreatic carcinoma | 2 months
  Vascularization parameters of pancreatic carcinoma:
  * on the primary tumor assessed by contrast-enhanced harmonic endoscopic ultrasonography (EUS)
  * and on liver metastases assessed by contrast enhanced ultrasonography (ceUS)

SECONDARY OUTCOMES:
Stiffness | 2 months
  Stiffness will be assessed in the primary tumor using ratio-elastography
Density | 2 months
  Density will be assessed in liver metastases on CTscan using density measurement before injection of contrast agent and after injection during the portal phase (80 sec post IV)
Safety | 2 months
  Adverse events of the treatment will be evaluated according to the Common Toxicity Criteria for Adverse Events (CTCAE version 4.03)
Response rate | 2 months
  Response rate will be evaluated according to RECIST V1.1 and CHOI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc RAOUL, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr/